CLINICAL TRIAL: NCT06622876
Title: Incidental Discovery of Pulmonary Emboli Via CT Scan: Impact of Detections on Patient Care and Resulting Complications. A Retrospective Study
Brief Title: Incidental Discovery of Pulmonary Emboli Via CT Scan: Impact of Detections on Patient Care and Resulting Complications
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: MMC-0216-24
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Computed tomography exam of the chest — Computed tomography exam of the chest done for other indications other than pulmonary emboli, in which incidental pulmonary embolism was detected.

SUMMARY:
In recent years, with an increase in the frequency of CT examinations, there has also been an increase in the random discovery of pulmonary emboli, often small, as part of examinations performed for other indications. Most of the literature so far deals with the discovery of such findings mainly in oncological patients, and there is relatively little information regarding the frequency of such random discovery in other patient populations. Specifically in the intensive care patient population, we have not yet found any study that examined the detection rates of these findings. Also, there is no consensus regarding how these random findings should be treated from a therapeutic point of view (whether to start treatment with full anticoagulation, and if so, for what period of time).

Random pulmonary embolism is often discovered as part of a CT scan done to assess acute lung disease or lung cancer staging. In a study done in oncology patients, 385 chest CT examinations were examined, with a random discovery of pulmonary emboli at a rate of 2.6% . A larger analysis of 8 studies involving 8491 cancer patients found a slightly higher incidence of 3.6%.

We would like to check the rate of pulmonary emboli that were randomly discovered in chest CT examinations performed in the intensive care unit for other indications, and the consequences of discoveries - ie starting anti-coagulant treatment and whether there were any complications for starting such treatment (bleeding).

ELIGIBILITY:
Inclusion Criteria: All patients who were admitted to the ICU between 8/2020 and 8/2024 and underwent chest CT during ICU stay -

Exclusion Criteria: Missing information

-

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who were admitted to the ICU between 8/2020 and 8/2024 and underwent chest CT during ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of incidental pulmonary embolism and related therapeutic consequences | 1.8.2020 - 1.8.2024
  To determine the rate of incidental pulmonary emboli that were discovered randomly in a CT scan in the intensive care unit and in what percentage of cases the findings caused a change in the patient's drug treatment (starting full anticoagulation therapy ).

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided